CLINICAL TRIAL: NCT06299579
Title: Phase III Clinical Trial of GD-11 for Injection in the Treatment of Acute Ischemic Stroke
Brief Title: GD-11 for Injection in the Treatment of Acute Ischemic Stroke
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Jiangsu Wangao Pharmaceutical Co. ltd (Unknown)
Responsible Party: Principal Investigator, Yongjun Wang, Chief Physician, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WG-GD11-III-01
Record Dates: First submitted 2024-02-27; First posted 2024-03-08 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Acute Ischemic Stroke
Keywords: Subjects within 48 hours
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: This trial is designed as a multicenter, randomized, double-blind, placebo-parallel controlled trial using a multicenter, randomized, double-blind, placebo-parallel controlled trial design. Subjects are randomly assigned in a 1:1 ratio and random number tables are generated using SAS（Statistics Analysis System）software.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GD-11 for injection test group (Experimental): GD-11 for injection, freeze-dried powder, 80mg, 160mg/dose Before the test drug is used, from the specification of 100 ml saline infusion bag, use a sterile syringe to extract about 15 ml saline into the test drug, by the oscillator or artificial vibration for about 5min, completely dissolved and then injected back to the administration of the infusion bag with a sterile syringe, gently shaking and mixing, and then intravenously titrated for 30min ± 10min.
  The first dose should be completed as soon as possible after randomization; the second dose should not be less than 6 hours from the start of the first dose, but not more than 12 + 1h; each subsequent dose interval of 12 ± 1h (calculated using the fixed time of administration as the baseline point and each dose should not be less than 6 hours from the start of the last dose); 10 consecutive days of treatment, a total of 20 times.
  Interventions: Drug: GD-11 for injection test group
- Placebo control group (Placebo Comparator): Placebo, freeze-dried powder, 80mg, 160mg/dose Before the test drug is used, from the specification of 100 ml saline infusion bag, use a sterile syringe to extract about 15 ml saline into the test drug, by the oscillator or artificial vibration for about 5min, completely dissolved and then injected back to the administration of the infusion bag with a sterile syringe, gently shaking and mixing, and then intravenously titrated for 30min ± 10min.
  The first dose should be completed as soon as possible after randomization; the second dose should not be less than 6 hours from the start of the first dose, but not more than 12 + 1h; each subsequent dose interval of 12 ± 1h (calculated using the fixed time of administration as the baseline point and each dose should not be less than 6 hours from the start of the last dose); 10 consecutive days of treatment, a total of 20 times.
  Interventions: Drug: Placebo control group

INTERVENTIONS:
Drug: GD-11 for injection test group — The first dose of GD-11 was administered as soon as possible after randomization and then every 12±1 hour. A total of 20 doses were required.
  Arms: GD-11 for injection test group
Drug: Placebo control group — The first dose of placebo was administered as soon as possible after randomization and then every 12±1 hour. A total of 20 doses were required.
  Arms: Placebo control group

SUMMARY:
Phase III Clinical Trial of GD-11 for Injection in the Treatment of Acute Ischemic Stroke - A Multi-Center, Randomized, Double-Blind, Parallel, Placebo-Controlled Phase III Clinical Study with the primary objective of evaluation of the efficacy and safety of GD-11 for injection in the treatment of acute ischemic stroke patients within 48 hours. The subject has a clinical diagnosis of acute ischemic stroke, within 48 hours from stroke onset to start of study treatment, with a National Institutes of Health Stroke Scale (NIHSS) between 6 and 20, had a total score of upper and lower limbs on motor deficits ≥ 2. The primary outcome is the proportion of subjects with mRS score ≤ 1 at 90 days after treatment.

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, parallel, placebo-controlled trial design was used. Subjects were randomly assigned in a 1:1 ratio to the experimental group (GD-11 for injection treatment group) and the control group (GD-11 for injection placebo group). Randomization stratification factors included onset time (≤24 hours, >24 hours) and center.Continuous treatment was performed for 10 days (20 times), followed up to 90 days after the first administration.

The trial was divided into three phases: screening/baseline phase, treatment phase, and follow-up phase.

Screening/baseline phase: Subjects entered the screening/baseline phase after signing the informed consent for screening examinations.

Treatment phase: Eligible subjects were randomly assigned in a 1:1 ratio to receive GD-11 for injection or placebo for injection for 10 days (20 times). During the treatment, protocol-required examinations were performed and safety was evaluated.

Follow-up phase: Subjects who completed the treatment entered the follow-up phase and were followed up to 90 days after the first administration.

Stroke-related scale scores were performed on the 10th, 30th, and 90th days after the first use of the test drug. Adverse events were recorded during the treatment and follow-up phases to further evaluate safety.

ELIGIBILITY:
Inclusion Criteria:

Only those who meet all of the following items will be enrolled:

1. age ≥18 years and <81 years, male or female;
2. National Institutes of Health Stroke Scale (NIHSS) score: 6 ≤ NIHSS ≤ 20, and the sum of item 5 Upper Extremity and item 6 Lower Extremity scores ≥ 2 after the onset of this event;
3. The onset of the disease is within 48 hours (including 48 hours);
4. Patients who are diagnosed with ischemic stroke according to the requirements of the latest guidelines such as "Diagnostic Points of Various Major Cerebrovascular Diseases in China 2019" or "Clinical Management Guidelines of Cerebrovascular Diseases in China (2nd edition)", and who have a good healing after the first onset or the last onset (mRS score ≤1 before this onset);
5. Obtaining informed consent approved by the Ethics Committee voluntarily signed by the patients or their legal representatives.

Exclusion Criteria:

Those who met one of the following items at screening will not be eligible for enrollment:

1. intracranial hemorrhagic disease as seen on cranial imaging: hemorrhagic stroke, epidural hematoma, intracranial hematoma, ventricular hemorrhage, subarachnoid hemorrhage, etc.; if blood seepage only, the suitability for enrollment may be based on the investigator's judgment;
2. severe impairment of consciousness: item score >1 on the 1a level of consciousness of the NIHSS;
3. thrombolysis, thrombolysis or intervention has been applied or is planned to be applied after this episode;
4. transient ischemic attack (TIA);
5. the patient's blood pressure remains ≥ 220 mmHg systolic or ≥ 120 mmHg diastolic after control;
6. patients with a previous diagnosis of severe mental disorders as well as patients with dementia;
7. patients who have been diagnosed with severe active liver disease, such as acute hepatitis, chronic active hepatitis, cirrhosis, etc.; or ALT (Alanine amino Transferase) or AST (Aspartate amino Transferase) > 2.0 x ULN (Upper Limit of Normal Value);
8. patients who have been diagnosed with severe active renal disease, renal insufficiency; or serum creatinine > 1.5 × ULN;
9. after the onset of the disease, the drug with neuroprotective effect has been used in the marketing, such as commercially available edaravone, edaravone dextran edaravone/(+)-2-Decanol injection concentrated solution, nimodipine, gangliosides, cytidine diphosphate, piracetam, oxiracetam, butylphenyl peptide, human urinary kallidinogenase (Urinary Kallidinogenase), cinepazide, murine nerve growth factor, cerebral vivax (hydrolysate of cerebral proteins), calf's blood deprivation of protein injection, calf's blood deprivation of protein extract injection and so on.
10. previously diagnosed with concurrent malignant tumors and undergoing anti-tumor therapy; for subjects diagnosed with malignant tumors after enrollment, continued participation in the study may be based on the investigator's judgment and the subject's wishes;
11. previously diagnosed with a serious systemic disease with an expected survival of <90 days;
12. the patient is pregnant, breastfeeding and the patient/patient's partner has the potential for pregnancy and plans to become pregnant during the trial period
13. patients with a previously known hypersensitivity to GD-11 for Injection and its excipients;
14. history of major surgery within 4 weeks prior to enrollment that in the investigator's assessment affects neurologic function scores or affects 90-day survival;
15. participation in another clinical study within 30 days prior to randomization or ongoing participation in another clinical study; Not considered by the investigator to be suitable for participation in this clinical study.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 980 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-02-22 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with mRS score ≤1 on 90th day of treatment | on 90th day of treatment
  Proportion of subjects with mRS score ≤1 on 90th day of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shuya Li, Study Director — IRB of Beijing Tiantan Hospital Capital Medical University Beijing
Locations (2):
- China (2):
  - Beijing Tiantan Hospital Capital Medical University Beijing, Beijing, Beijing Municipality
  - Linfen Central Hospital, Shangxi, Linfen City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Motwani JG, Lipworth BJ. Clinical pharmacokinetics of drug administered buccally and sublingually. Clin Pharmacokinet. 1991 Aug;21(2):83-94. doi: 10.2165/00003088-199121020-00001. No abstract available. PMID 1884569
- [Result] Sato T, Mizuno K, Ishii F. A novel administration route of edaravone--II: mucosal absorption of edaravone from edaravone/hydroxypropyl-beta-cyclodextrin complex solution including L-cysteine and sodium hydrogen sulfite. Pharmacology. 2010;85(2):88-94. doi: 10.1159/000276548. Epub 2010 Jan 21. PMID 20110753
- [Result] Enlimomab Acute Stroke Trial Investigators. Use of anti-ICAM-1 therapy in ischemic stroke: results of the Enlimomab Acute Stroke Trial. Neurology. 2001 Oct 23;57(8):1428-34. doi: 10.1212/wnl.57.8.1428. PMID 11673584
- [Result] Cui L, Hung HM, Wang SJ. Modification of sample size in group sequential clinical trials. Biometrics. 1999 Sep;55(3):853-7. doi: 10.1111/j.0006-341x.1999.00853.x. PMID 11315017
- [Result] Mehta CR, Pocock SJ. Adaptive increase in sample size when interim results are promising: a practical guide with examples. Stat Med. 2011 Dec 10;30(28):3267-84. doi: 10.1002/sim.4102. Epub 2010 Nov 30. PMID 22105690